CLINICAL TRIAL: NCT04211948
Title: Prospective Cohort Study Comparing Robotic and Open Surgery for Pancreatic Cancer
Brief Title: Clinical Study Between Robotic and Open Surgery in Patients With Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kai Qin, Principal Investigator, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HBP-RWR-001
Record Dates: First submitted 2019-11-29; First posted 2019-12-26 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Minimally Invasive Surgery
Keywords: Robotic assisted surgery
MeSH Terms: interventions — Robotic Surgical Procedures; Conversion to Open Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robotic pancreatectomy (Experimental): robotic pancreatectomy(including pancreaticoduodenectomy and distal pancreatectomy)
  Interventions: Procedure: robotic surgery
- open surgery (Active Comparator): open pancreatectomy(including pancreaticoduodenectomy and distal pancreatectomy)
  Interventions: Procedure: open surgery

INTERVENTIONS:
Procedure: robotic surgery — Pancreatectomy with robotic assisted system
  Arms: robotic pancreatectomy
Procedure: open surgery — Traditional open pancreatectomy
  Arms: open surgery

SUMMARY:
The purpose of this study is to determine whether robotic surgery has limitations in terms of patient age, tumor size, location, and vascular relationship when compared to open surgery for pancreatic cancer. Whether robotic surgery has advantages over intraoperative bleeding, operative time, postoperative complications (bleeding, infection, pancreatic fistula) and postoperative hospital stays compared to open surgery.And the differences in lymph nodes harvest and postoperative survival between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed pancreatic ductal adenocarcinoma
* Patients and their families volunteered to test and signed informed consent.

Exclusion Criteria:

* Preoperative exclusion:

  1. Patients with metastasis (M1)
  2. Patients with tumor recurrence
  3. Patients with artery and/or vein invasion and can't perform radical resection and reconstruction
  4. Patients with poor cardiopulmonary function cannot tolerate surgery;
  5. receive neoadjuvant radiotherapy and chemotherapy before surgery;
  6. The patient or family member refuses to join the group;
  7. Pregnant patients
* Intraoperative exclusion:

  1. Intraoperative exploration of metastases in other parts besides the primary lesion
  2. Other organs malignant tumors metastasize to the pancreas
* Postoperative exclusion:

  1. pathology confirmed non-pancreatic ductal adenocarcinoma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
1 year overall survival rate | 1 year post-operation
3 years overall survival rate | 3 years post-operation

SECONDARY OUTCOMES:
Postoperative Complications | Within 90 days or before discharge
  pancreatic fistula, bile leakage, hemorrhage, DGE, etc
1, 3years disease free survival rate | 1,3years post-operation

CONTACTS AND LOCATIONS:
Overall Officials: Kai Qin, Principal Investigator — Ruijin Hospital
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No